CLINICAL TRIAL: NCT00581074
Title: Effects of Grapefruit or Grapefruit Juice on Anthropometry, Dietary Intakes, Appetite, and Metabolic Profile in Overweight and Obese Young and Middle-Aged Adults
Acronym: GJW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Heidi J. Silver, State of Florida Dept of Citrus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 060035
Record Dates: First submitted 2007-12-17; First posted 2007-12-27 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Obesity
Keywords: obesity; diet; weight loss; metabolic syndrome
MeSH Terms: conditions — Obesity; Weight Loss; Metabolic Syndrome | interventions — Diet; grapefruit seed extract

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- G (Active Comparator): grapefruit
  Interventions: Behavioral: diet (grapefruit or grapefruit juice)
- J (Active Comparator): Juice
  Interventions: Behavioral: diet (grapefruit or grapefruit juice)
- W (Placebo Comparator): placebo
  Interventions: Behavioral: diet (grapefruit or grapefruit juice)

INTERVENTIONS:
Behavioral: diet (grapefruit or grapefruit juice) — weight loss diet

SUMMARY:
This trial examines the effects of grapefruit or grapefruit juice on anthropometry, dietary intakes, appetite, and metabolic profile in overweight and obese young and middle-aged adults.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-39.9

Exclusion Criteria:

* Pregnant or lactating
* On medications that are interfered with by consuming grapefruit juice

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
weight loss | 3 months

SECONDARY OUTCOMES:
metabolic syndrome | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Heidi J Silver, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Silver HJ, Dietrich MS, Niswender KD. Effects of grapefruit, grapefruit juice and water preloads on energy balance, weight loss, body composition, and cardiometabolic risk in free-living obese adults. Nutr Metab (Lond). 2011 Feb 2;8(1):8. doi: 10.1186/1743-7075-8-8. PMID 21288350